CLINICAL TRIAL: NCT05059080
Title: A Multicenter, Observational, 6-Month Follow-up Study of Patients With COVID-19 Previously Enrolled in a RO7496998 (AT-527) Study
Brief Title: A Six-Month Follow-Up Study of Participants With Coronavirus Disease 2019 (COVID-19) Previously Enrolled in a RO7496998 (AT-527) Study
Acronym: MEADOWSPRING
Status: Terminated | Type: Observational
Why Stopped: Based on program revaluation and in agreement with the co-development partner the sponsor took the decision to terminate this study.
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Atea Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CV43140; 2021-000627-12 (EudraCT Number)
Record Dates: First submitted 2021-09-24; First posted 2021-09-28 (Actual); Results first posted 2023-07-28 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2022-09

CONDITIONS: COVID-19; Long COVID
Keywords: Coronavirus Disease 2019; COVID-19; SARS-CoV-2; Mild to Moderate COVID-19; Long-COVID; Observational
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants Diagnosed with COVID-19: Participants were previously enrolled in a RO7496998 (AT-527) study (i.e. parent study NCT04889040 [CV43043]).

SUMMARY:
This study will evaluate the long-term sequelae of COVID-19 in patients diagnosed with COVID-19 who previously enrolled in a RO7496998 (AT-527) study (i.e. parent study NCT04889040 [CV43043]), for approximately 6 months after the end of the parent study.

ELIGIBILITY:
Inclusion Criteria:

* Participant was diagnosed with COVID-19 and enrolled in a Phase III RO7496998 (AT-527) COVID-19 study

Exclusion Criteria:

* Participation in an interventional study at the time of enrollment or plans to enroll in an interventional study during this study.
* Any serious medical condition or abnormality of clinical laboratory tests that, in the investigator's judgment, precludes the patient's safe participation in and completion of the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants enrolled in a RO7496998 (AT-527) study.
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2022-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (35):
- Instituto Ave Pulmo, Mar del Plata, Argentina
- Belgium (2):
  - Private Practice Dr Jean Benoit Martinot, Erpent
  - Medif, Gozée
- Brazil (5):
  - L2IP -Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - Chronos Pesquisa Clinica, Taguatinga, Federal District
  - Hospital Nossa Senhora das Graças, Curitiba, Paraná
  - Hospital Agamenon Magalhães, Recife, Pernambuco
  - Conjunto Hospitalar do Mandaqui, São Paulo, São Paulo
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet Copenhagen University Hospital, Copenhagen
  - Sjællands Universitetshospital, Roskilde, Roskilde
- Praxis am Ebertplatz, Cologne, Germany
- Mexico (6):
  - CIMAB SA de CV, Torreón, Coahuila
  - Panamerican Clinical Research S.A de C.V., Guadalajara, Jalisco
  - Clinstile S.A de C.V., Mexico City, Mexico CITY (federal District)
  - PanAmerican Clinical Research, Querétaro, Queréaro, Querétaro
  - Instituto Jalisciense de Investigacion Clinica S.A. de C.V., Guadalajara
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, México
- Romania (3):
  - Prof. Dr. Matei Bals Institute of Infectious Diseases, Bucharest
  - County Hospital Caracal, Caracal
  - Sibiu Emergency Clinical County Hospital, Sibiu
- Universitätsspital Zürich, Zurich, Switzerland
- Turkey (Türkiye) (5):
  - Gazi Universitesi Tip Fakultesi, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Ankara University Medical Faculty - PPDS, Çankaya
  - Ege University Medical Faculty, Izmir
  - Karadeniz Technical University Faculty of Medicine, Trabzon
- Ukraine (8):
  - Municipal Non-profit enterprise Central City Clinical Hospital of Ivano-Frankivsk City Council, Ivano-Frankivsk, Katerynoslav Governorate
  - Municipal Non-profit Enterprise "City Clinical Hospital #13" of Kharkiv City Council, Kharkiv, Kharkiv Governorate
  - CNPE City Clinical Hospital #6 of DCC, Dnipro, Kholm Governorate
  - Medical Center LLC "Harmony of Beauty", Kyiv, KIEV Governorate
  - CNE Kyiv City Clinical Hospital#1 of Exec. Body, Kyiv, KIEV Governorate
  - Kyiv Railway Clinical Hospital No2 of Branch Health Center of the JSC Ukrainian Rail, Kyiv, KIEV Governorate
  - Communal Non-Commercial Enterprise Vinnytsia City Clinical Hospital 1, Vinnytsia, Podolia Governorate
  - Communal Non-Profit Enterprise City Hospital #7 of Zaporizhzhia City Council, Zaporizhzhia, Tavria Okruha

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants diagnosed with COVID-19, who previously enrolled in a RO7496998 (AT-527) study (i.e. parent study NCT04889040 [CV43043]), were enrolled in this study after the end of the parent study.
Groups:
- All Participants: Participants were previously enrolled in a RO7496998 (AT-527) study (i.e. parent study NCT04889040 [CV43043]).
Period: Overall Study
Arm/Group | All Participants
Started | 72
Completed | 5
Not Completed | 67
Not completed — Withdrawal by Subject | 3
Not completed — Study Terminated by Sponsor | 64

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43
  Male | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 51
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 12
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Percentage of Participants With COVID-19 Symptoms Assessed through the COVID-19 Symptom Diary [Number; unit: percentage of participants] — The COVID-19 Symptom Diary included the following 14 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, diarrhea, sense of smell over the past 7 days, sense of taste over the past 7 days. Reported here is the percentage of participants for the following: items 1-12 = mild-severe; items 13-14 = less than usual OR no sense of smell/taste. Baseline is approximately one month after the initial infection. Population: For the study-specific baseline characteristic the number of participants indicates participants with data available for analysis at baseline.
  percentage of participants
    Nasal Congestion or Runny Nose: number analyzed (Participants) | 69
    Nasal Congestion or Runny Nose | 17.4
    Sore Throat: number analyzed (Participants) | 69
    Sore Throat | 7.2
    Cough: number analyzed (Participants) | 69
    Cough | 21.7
    Shortness of Breath: number analyzed (Participants) | 69
    Shortness of Breath | 5.8
    Muscle or Body Aches: number analyzed (Participants) | 69
    Muscle or Body Aches | 21.7
    Fatigue: number analyzed (Participants) | 69
    Fatigue | 31.9
    Headache: number analyzed (Participants) | 69
    Headache | 13.0
    Chills/Sweats: number analyzed (Participants) | 69
    Chills/Sweats | 5.8
    Feeling Hot or Feverish: number analyzed (Participants) | 69
    Feeling Hot or Feverish | 4.3
    Nausea: number analyzed (Participants) | 69
    Nausea | 4.3
    Vomiting: number analyzed (Participants) | 69
    Vomiting | 0
    Diarrhea: number analyzed (Participants) | 69
    Diarrhea | 2.9
    Reduction or Loss of Sense of Smell over the Past 7 Days: number analyzed (Participants) | 69
    Reduction or Loss of Sense of Smell over the Past 7 Days | 23.2
    Reduction or Loss of Sense of Taste over the Past 7 Days: number analyzed (Participants) | 69
    Reduction or Loss of Sense of Taste over the Past 7 Days | 17.4

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With COVID-19 Symptoms Assessed Through the COVID-19 Symptom Diary up to Month 6
Description: COVID-19 symptoms were evaluated using the COVID-19 Symptom Diary. The COVID-19 Symptom Diary included the following 14 items: nasal congestion or runny nose, sore throat, cough, shortness of breath, muscle or body aches, fatigue, headache, chills/sweats, feeling hot or feverish, nausea, vomiting, diarrhea, sense of smell over the past 7 days and sense of taste over the past 7 days. The severity of items 1-12 were recorded on a 4-point Likert scale (i.e none/mild/moderate/severe). Items 13-14 were recorded on a 3-point Likert scale (i.e. same as usual/less than usual/no sense). Reported here is the percentage of participants with COVID-19 symptoms (mild/moderate/severe or less than usual/no sense) recorded during week 4 of each month following the baseline assessment.
Time Frame: Month 1 - Week 4, Month 2 - Week 4, Month 3 - Week 4, Month 4 - Week 4, Month 5 - Week 4, Month 6 - Week 4
Population: The analysis population included all participants enrolled in the study. The number of participants analyzed at each time point includes all participants with data available for the specific time point. All enrolled participants contributed to the outcome measure results.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants
  Nasal Congestion or Runny Nose: Month 1 - Week 4: number analyzed (Participants) | 61
  Nasal Congestion or Runny Nose: Month 1 - Week 4 | 18.0
  Nasal Congestion or Runny Nose: Month 2 - Week 4: number analyzed (Participants) | 64
  Nasal Congestion or Runny Nose: Month 2 - Week 4 | 17.2
  Nasal Congestion or Runny Nose: Month 3 - Week 4: number analyzed (Participants) | 59
  Nasal Congestion or Runny Nose: Month 3 - Week 4 | 18.6
  Nasal Congestion or Runny Nose: Month 4 - Week 4: number analyzed (Participants) | 32
  Nasal Congestion or Runny Nose: Month 4 - Week 4 | 15.6
  Nasal Congestion or Runny Nose: Month 5 - Week 4: number analyzed (Participants) | 14
  Nasal Congestion or Runny Nose: Month 5 - Week 4 | 21.4
  Nasal Congestion or Runny Nose: Month 6 - Week 4: number analyzed (Participants) | 3
  Nasal Congestion or Runny Nose: Month 6 - Week 4 | 0
  Sore Throat: Month 1 - Week 4: number analyzed (Participants) | 61
  Sore Throat: Month 1 - Week 4 | 9.8
  Sore Throat: Month 2 - Week 4: number analyzed (Participants) | 64
  Sore Throat: Month 2 - Week 4 | 14.1
  Sore Throat: Month 3 - Week 4: number analyzed (Participants) | 59
  Sore Throat: Month 3 - Week 4 | 15.3
  Sore Throat: Month 4 - Week 4: number analyzed (Participants) | 32
  Sore Throat: Month 4 - Week 4 | 18.8
  Sore Throat: Month 5 - Week 4: number analyzed (Participants) | 14
  Sore Throat: Month 5 - Week 4 | 0
  Sore Throat: Month 6 - Week 4: number analyzed (Participants) | 3
  Sore Throat: Month 6 - Week 4 | 0
  Cough: Month 1 - Week 4: number analyzed (Participants) | 61
  Cough: Month 1 - Week 4 | 16.4
  Cough: Month 2 - Week 4: number analyzed (Participants) | 64
  Cough: Month 2 - Week 4 | 17.2
  Cough: Month 3 - Week 4: number analyzed (Participants) | 59
  Cough: Month 3 - Week 4 | 16.9
  Cough: Month 4 - Week 4: number analyzed (Participants) | 32
  Cough: Month 4 - Week 4 | 15.6
  Cough: Month 5 - Week 4: number analyzed (Participants) | 14
  Cough: Month 5 - Week 4 | 7.1
  Cough: Month 6 - Week 4: number analyzed (Participants) | 3
  Cough: Month 6 - Week 4 | 0
  Shortness of Breath: Month 1 - Week 4: number analyzed (Participants) | 61
  Shortness of Breath: Month 1 - Week 4 | 11.5
  Shortness of Breath: Month 2 - Week 4: number analyzed (Participants) | 64
  Shortness of Breath: Month 2 - Week 4 | 12.5
  Shortness of Breath: Month 3 - Week 4: number analyzed (Participants) | 59
  Shortness of Breath: Month 3 - Week 4 | 18.6
  Shortness of Breath: Month 4 - Week 4: number analyzed (Participants) | 32
  Shortness of Breath: Month 4 - Week 4 | 12.5
  Shortness of Breath: Month 5 - Week 4: number analyzed (Participants) | 14
  Shortness of Breath: Month 5 - Week 4 | 7.1
  Shortness of Breath: Month 6 - Week 4: number analyzed (Participants) | 3
  Shortness of Breath: Month 6 - Week 4 | 0
  Muscle or Body Aches: Month 1 - Week 4: number analyzed (Participants) | 61
  Muscle or Body Aches: Month 1 - Week 4 | 13.1
  Muscle or Body Aches: Month 2 - Week 4: number analyzed (Participants) | 64
  Muscle or Body Aches: Month 2 - Week 4 | 18.8
  Muscle or Body Aches: Month 3 - Week 4: number analyzed (Participants) | 59
  Muscle or Body Aches: Month 3 - Week 4 | 18.6
  Muscle or Body Aches: Month 4 - Week 4: number analyzed (Participants) | 32
  Muscle or Body Aches: Month 4 - Week 4 | 12.5
  Muscle or Body Aches: Month 5 - Week 4: number analyzed (Participants) | 14
  Muscle or Body Aches: Month 5 - Week 4 | 14.3
  Muscle or Body Aches: Month 6 - Week 4: number analyzed (Participants) | 3
  Muscle or Body Aches: Month 6 - Week 4 | 0
  Fatigue: Month 1 - Week 4: number analyzed (Participants) | 61
  Fatigue: Month 1 - Week 4 | 27.9
  Fatigue: Month 2 - Week 4: number analyzed (Participants) | 64
  Fatigue: Month 2 - Week 4 | 26.6
  Fatigue: Month 3 - Week 4: number analyzed (Participants) | 59
  Fatigue: Month 3 - Week 4 | 35.6
  Fatigue: Month 4 - Week 4: number analyzed (Participants) | 32
  Fatigue: Month 4 - Week 4 | 25.0
  Fatigue: Month 5 - Week 4: number analyzed (Participants) | 14
  Fatigue: Month 5 - Week 4 | 28.6
  Fatigue: Month 6 - Week 4: number analyzed (Participants) | 3
  Fatigue: Month 6 - Week 4 | 0
  Headache: Month 1 - Week 4: number analyzed (Participants) | 61
  Headache: Month 1 - Week 4 | 6.6
  Headache: Month 2 - Week 4: number analyzed (Participants) | 64
  Headache: Month 2 - Week 4 | 7.8
  Headache: Month 3 - Week 4: number analyzed (Participants) | 59
  Headache: Month 3 - Week 4 | 20.3
  Headache: Month 4 - Week 4: number analyzed (Participants) | 32
  Headache: Month 4 - Week 4 | 12.5
  Headache: Month 5 - Week 4: number analyzed (Participants) | 14
  Headache: Month 5 - Week 4 | 0
  Headache: Month 6 - Week 4: number analyzed (Participants) | 3
  Headache: Month 6 - Week 4 | 0
  Chills/Sweats: Month 1 - Week 4: number analyzed (Participants) | 61
  Chills/Sweats: Month 1 - Week 4 | 0
  Chills/Sweats: Month 2 - Week 4: number analyzed (Participants) | 64
  Chills/Sweats: Month 2 - Week 4 | 7.8
  Chills/Sweats: Month 3 - Week 4: number analyzed (Participants) | 59
  Chills/Sweats: Month 3 - Week 4 | 6.8
  Chills/Sweats: Month 4 - Week 4: number analyzed (Participants) | 32
  Chills/Sweats: Month 4 - Week 4 | 6.3
  Chills/Sweats: Month 5 - Week 4: number analyzed (Participants) | 14
  Chills/Sweats: Month 5 - Week 4 | 0
  Chills/Sweats: Month 6 - Week 4: number analyzed (Participants) | 3
  Chills/Sweats: Month 6 - Week 4 | 0
  Feeling Hot or Feverish: Month 1 - Week 4: number analyzed (Participants) | 61
  Feeling Hot or Feverish: Month 1 - Week 4 | 3.3
  Feeling Hot or Feverish: Month 2 - Week 4: number analyzed (Participants) | 64
  Feeling Hot or Feverish: Month 2 - Week 4 | 6.3
  Feeling Hot or Feverish: Month 3 - Week 4: number analyzed (Participants) | 59
  Feeling Hot or Feverish: Month 3 - Week 4 | 5.1
  Feeling Hot or Feverish: Month 4 - Week 4: number analyzed (Participants) | 32
  Feeling Hot or Feverish: Month 4 - Week 4 | 3.1
  Feeling Hot or Feverish: Month 5 - Week 4: number analyzed (Participants) | 14
  Feeling Hot or Feverish: Month 5 - Week 4 | 0
  Feeling Hot or Feverish: Month 6 - Week 4: number analyzed (Participants) | 3
  Feeling Hot or Feverish: Month 6 - Week 4 | 0
  Nausea: Month 1 - Week 4: number analyzed (Participants) | 61
  Nausea: Month 1 - Week 4 | 0
  Nausea: Month 2 - Week 4: number analyzed (Participants) | 64
  Nausea: Month 2 - Week 4 | 6.3
  Nausea: Month 3 - Week 4: number analyzed (Participants) | 59
  Nausea: Month 3 - Week 4 | 10.2
  Nausea: Month 4 - Week 4: number analyzed (Participants) | 32
  Nausea: Month 4 - Week 4 | 6.3
  Nausea: Month 5 - Week 4: number analyzed (Participants) | 14
  Nausea: Month 5 - Week 4 | 0
  Nausea: Month 6 - Week 4: number analyzed (Participants) | 3
  Nausea: Month 6 - Week 4 | 0
  Vomiting: Month 1 - Week 4: number analyzed (Participants) | 61
  Vomiting: Month 1 - Week 4 | 0
  Vomiting: Month 2 - Week 4: number analyzed (Participants) | 64
  Vomiting: Month 2 - Week 4 | 1.6
  Vomiting: Month 3 - Week 4: number analyzed (Participants) | 59
  Vomiting: Month 3 - Week 4 | 3.4
  Vomiting: Month 4 - Week 4: number analyzed (Participants) | 32
  Vomiting: Month 4 - Week 4 | 0
  Vomiting: Month 5 - Week 4: number analyzed (Participants) | 14
  Vomiting: Month 5 - Week 4 | 0
  Vomiting: Month 6 - Week 4: number analyzed (Participants) | 3
  Vomiting: Month 6 - Week 4 | 0
  Diarrhea: Month 1 - Week 4: number analyzed (Participants) | 61
  Diarrhea: Month 1 - Week 4 | 1.6
  Diarrhea: Month 2 - Week 4: number analyzed (Participants) | 64
  Diarrhea: Month 2 - Week 4 | 4.7
  Diarrhea: Month 3 - Week 4: number analyzed (Participants) | 59
  Diarrhea: Month 3 - Week 4 | 5.1
  Diarrhea: Month 4 - Week 4: number analyzed (Participants) | 32
  Diarrhea: Month 4 - Week 4 | 9.4
  Diarrhea: Month 5 - Week 4: number analyzed (Participants) | 14
  Diarrhea: Month 5 - Week 4 | 0
  Diarrhea: Month 6 - Week 4: number analyzed (Participants) | 3
  Diarrhea: Month 6 - Week 4 | 0
  Reduction of Loss of Sense of Smell over the Past 7 Days: Month 1 - Week 4: number analyzed (Participants) | 61
  Reduction of Loss of Sense of Smell over the Past 7 Days: Month 1 - Week 4 | 18.0
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 2 - Week 4: number analyzed (Participants) | 64
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 2 - Week 4 | 18.8
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 3 - Week 4: number analyzed (Participants) | 59
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 3 - Week 4 | 18.6
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 4 - Week 4: number analyzed (Participants) | 32
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 4 - Week 4 | 15.6
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 5 - Week 4: number analyzed (Participants) | 14
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 5 - Week 4 | 21.4
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 6 - Week 4: number analyzed (Participants) | 3
  Reduction or Loss of Sense of Smell over the Past 7 Days: Month 6 - Week 4 | 0
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 1 - Week 4: number analyzed (Participants) | 61
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 1 - Week 4 | 11.5
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 2 - Week 4: number analyzed (Participants) | 64
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 2 - Week 4 | 15.6
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 3 - Week 4: number analyzed (Participants) | 59
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 3 - Week 4 | 13.6
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 4 - Week 4: number analyzed (Participants) | 32
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 4 - Week 4 | 15.6
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 5 - Week 4: number analyzed (Participants) | 14
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 5 - Week 4 | 21.4
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 6 - Week 4: number analyzed (Participants) | 3
  Reduction or Loss of Sense of Taste over the Past 7 Days: Month 6 - Week 4 | 0

2. Secondary Outcome: Dyspnea Symptoms Assessment Score Through the Patient Reported Outcomes Measurement Information System - Short Form (PROMIS-SF) - Dyspnea Questionnaire
Description: The PROMIS-SF-Dyspnea Questionnaire is a 10-item questionnaire to evaluate the impact of dyspnea on specific activities. Participants self-assessed the severity of shortness of breath and difficulty of breathing in response to specific activities with a recall of the past 7 days. The PROMIS SF-Dyspnea Severity instrument is scored on a 4-point Likert scale, with an option to indicate that an activity had not been performed. Total score range is 0-30, where a higher score indicates a higher symptom severity of dyspnea.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: The analysis population included all enrolled participants in the study for whom data were available at each time point as indicated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 72
score on a scale
  Baseline: number analyzed (Participants) | 70
  Baseline | 2.04 (3.62)
  Month 1: number analyzed (Participants) | 59
  Month 1 | 1.94 (3.49)
  Month 2: number analyzed (Participants) | 63
  Month 2 | 2.12 (3.69)
  Month 3: number analyzed (Participants) | 58
  Month 3 | 1.97 (2.97)
  Month 4: number analyzed (Participants) | 30
  Month 4 | 1.33 (2.95)
  Month 5: number analyzed (Participants) | 13
  Month 5 | 0.69 (1.70)
  Month 6: number analyzed (Participants) | 3
  Month 6 | 0.00 (0.00)

3. Secondary Outcome: Respiratory-specific Health-related Quality of Life Score as Assessed by the St. George's Respiratory Questionnaire (SGRQ)
Description: The SGRQ is a 50-item respiratory-specific health-related quality of life instrument that measures health impairment. The questionnaire contains 3 domains: symptoms, activity, and impacts. Items were assessed on various response scales, including a 5-point Likert scale and True/False scale. Each scale is scored from 0 to 100, and the total score represents the weighted average of these three subscores. Higher scores correspond to worse quality of life. The SGRQ had a recall specification of 4 weeks.
Time Frame: Baseline, Month 1, Month 2, Month 3, Month 4, Month 5, Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Participants
Number analyzed (Participants) | 72
score on a scale
  Baseline: number analyzed (Participants) | 70
  Baseline | 12.93 (16.57)
  Month 1: number analyzed (Participants) | 59
  Month 1 | 11.13 (16.27)
  Month 2: number analyzed (Participants) | 60
  Month 2 | 11.39 (16.35)
  Month 3: number analyzed (Participants) | 59
  Month 3 | 11.40 (16.27)
  Month 4: number analyzed (Participants) | 32
  Month 4 | 13.88 (23.91)
  Month 5: number analyzed (Participants) | 13
  Month 5 | 6.66 (14.70)
  Month 6: number analyzed (Participants) | 3
  Month 6 | 3.46 (4.11)

4. Secondary Outcome: Percentage of Participants With COVID-19 Related Medically-Attended Visits
Description: COVID-19-related medically-attended visits were defined as hospitalization, ER visit, urgent care visit, physician's office visit, or telemedicine visit with the primary reason for the visit being COVID-19 or COVID-19-related symptoms.
Time Frame: Up to 6 months
Population: The analysis population included all enrolled participants in the study.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants | 2.8 [0.00 to 7.81]

5. Secondary Outcome: Percentage of Participants With Death Attributable to Progression of COVID-19
Time Frame: Up to 6 months
Population: The analysis population included all enrolled participants in the study.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants | 0

6. Secondary Outcome: Percentage of Participants Re-Infected With Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2)
Description: Reinfection was defined as any nasopharyngeal (NP) swab that was positive for SARS-CoV-2 infection via reverse-transcriptase polymerase chain reaction (RT-PCR), taken when clinically indicated based on symptoms.
Time Frame: Up to 6 months
Population: The analysis population included all enrolled participants in the study.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants | 0

7. Secondary Outcome: Percentage of Participants With Any Post-Treatment Infection
Description: Post-treatment infections were defined as any adverse event with a primary system organ class of infections and infestations.
Time Frame: Up to 6 months
Population: The analysis population included all enrolled participants in the study.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants | 8.3 [0.34 to 16.33]

8. Secondary Outcome: Percentage of Participants With COVID-19-Related Complications
Description: COVID-19 related complications included pneumonia, acute respiratory failure, sepsis, coagulopathy, pericarditis and/or myocarditis, and cardiac failure.
Time Frame: Up to 6 months
Population: The analysis population included all enrolled participants in the study.
Measure: Number (97.5% Confidence Interval); unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants | 0 [0.00 to 0.69]

9. Secondary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a clinical investigation subject administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any of the following: any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the medicinal product, any new disease or exacerbation of an existing disease, recurrence of an intermittent medical condition not present at baseline or related to a protocol-mandated intervention.
Time Frame: Up to 6 months
Population: The safety population included all enrolled participants in the study.
Measure: Number; unit: percentage of participants
Arm/Group | All Participants
Number analyzed (Participants) | 72
percentage of participants | 26.4

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: All AEs/Serious AEs continuing/persisting from the parent study or any new AEs with an onset date on or after the first day of enrollment and during this follow-up study are displayed. The safety population included all participants enrolled in the study.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/72
Serious Adverse Events (participants affected / at risk) | 2/72
Other Adverse Events (participants affected / at risk) | 17/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=72)
Cataract (Eye disorders) | 1 (1)
Arterial occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=72)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1)
Chest discomfort (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hangover (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Vaccination site pain (General disorders) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Vaginal infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (3)
Hyposmia (Nervous system disorders) | 1 (1)
Taste disorder (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-03): https://cdn.clinicaltrials.gov/large-docs/80/NCT05059080/Prot_SAP_000.pdf